CLINICAL TRIAL: NCT03795831
Title: Validation Study in Patients of a Non-invasive Blood Pressure Monitor for Perioperative Use
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, D.P.Veelo, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2017-14
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Intraoperative Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cohort: Adult patients, undergoing surgery requiring general anesthesia, planned to be monitored with a system that accurately measures and stores the intra-arterial waveform.
  Interventions: Device: ClearSight feasibility testing

INTERVENTIONS:
Device: ClearSight feasibility testing — A cuff is placed on a finger of the patient. The ClearSight system uses a volume clamp technology allowing measuring of continuous blood pressure waveform. Note: There will only be observational recordings, no interventions

SUMMARY:
Collecting all available data (waveforms, beat to beat data, status data) generated by a non invasive blood pressure monitor on each hand and compare this to the actual data obtained by intra arterial (radial) monitoring.

This to see if the non invasive bloodpressure monitor can be validated for intraoperative use.

DETAILED DESCRIPTION:
Although a blood pressure monitoring device could be evaluated by the comparing systolic, diastolic and mean arterial pressure to a reference pressure, it is the specific aim to collect all available data (waveforms, beat to beat data, status data) generated by the blood pressure monitor.

After data analysis and comparison to patient's actual intra-arterial waveform, the outcome will be evaluated by Association for the Advancement of Medical Instrumentation (AAMI) standards to see if the non invasive bloodpressure monitor can be validated for intraoperative use.

The study is targeted at patients already monitored with a system that accurately measures and stores the intra-arterial waveform, such as the FloTrac system in the EV1000 monitor.

This study is a substudy of a feasability protocol evaluating a new algorithm for the Clearsight system.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose arterial blood pressure is measured invasively with technology that allows for the storage of the intra-arterial waveform with sufficient quality and resolution (Flotrac).
* Patients older than 18, for elective general surgery.

Exclusion Criteria:

- Patient conditions that are expected to potentially and significantly affect the transfer of pressure between radial artery and the finger, e.g. due to recent finger fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in a perioperative setting already monitored with a system that accurately measures and stores the intra-arterial waveform, such as the FloTrac system in the EV1000 monitor.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
validation systole, diastole, mean ABP and pulse pressure | within 1 hour
  accuracy and precision of invasive blood pressure curve vs non-invasive blood pressure curves(ipsilateral and contralateral)
implementation of software alterations to improve systole, diastole, mean ABP accuracy and pulse pressure | time during surgery
  Comparison of the non-invasive blood pressure curve after software alterations to the reference and invasive arterial blood pressure curve

CONTACTS AND LOCATIONS:
Overall Officials: D.P. Veelo, Dr, Principal Investigator — inverstigator
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rellum SR, Noteboom SH, van der Ster BJP, Schuurmans J, Kho E, Vlaar APJ, Schenk J, Veelo DP. The hypotension prediction index versus mean arterial pressure in predicting intraoperative hypotension: A clinical perspective. Eur J Anaesthesiol. 2025 Jun 1;42(6):527-535. doi: 10.1097/EJA.0000000000002150. Epub 2025 Feb 27. PMID 40012367
- [Derived] Rellum SR, Kho E, Schenk J, van der Ster BJP, Vlaar APJ, Veelo DP. A comparison between invasive and noninvasive measurement of the Hypotension Prediction Index: A post hoc analysis of a prospective cohort study. Eur J Anaesthesiol. 2025 Feb 1;42(2):131-139. doi: 10.1097/EJA.0000000000002082. Epub 2024 Oct 16. PMID 39411994
- [Derived] Kho E, van der Ster BJP, van der Ven WH, Vlaar APJ, Immink RV, Veelo DP. Clinical agreement of a novel algorithm to estimate radial artery blood pressure from the non-invasive finger blood pressure. J Clin Anesth. 2022 Dec;83:110976. doi: 10.1016/j.jclinane.2022.110976. Epub 2022 Sep 26. PMID 36174389